CLINICAL TRIAL: NCT00761137
Title: A Two-Phase, Double Blind, Placebo-Controlled, Randomized, Crossover Study of the Safety and Efficacy of Intra-Oral NH004 Films for the Short-Term Relief of Sialorrhea Symptoms in Parkinson's Disease Patients
Brief Title: Safety and Efficacy Study of NH004 Films for Relief of Sialorrhea Symptoms in Parkinson's Disease Patients
Acronym: NH004-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroHealing Pharmaceuticals Inc. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH004-2
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2013-04

CONDITIONS: Sialorrhea Secondary to Parkinson's Disease
Keywords: sialorrhea; drooling; excessive salivation; parkinson's disease
MeSH Terms: conditions — Sialorrhea; Parkinson Disease | interventions — Tropicamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tropicamide placebo (Experimental): subject received (blinded) each of the 4 drug doses at different visits - 0 mg tropicamide, 0.3 mg tropicamide, 1 mg tropicamide, 3 mg tropicamide
  Interventions: Drug: 0.3 mg tropicamide; Drug: 1 mg tropicamide; Drug: 3 mg tropicamide; Drug: 0 mg tropicamide
- Tropicamide 0.3 mg (Experimental): subject received (blinded) each of the 4 drug doses at different visits - 0.3 mg tropicamide, 1 mg tropicamide, 3 mg tropicamide, 0 mg tropicamide
  Interventions: Drug: 0.3 mg tropicamide; Drug: 1 mg tropicamide; Drug: 3 mg tropicamide; Drug: 0 mg tropicamide
- Tropicamide 1 mg (Experimental): subject received (blinded) each of the 4 drug doses at different visits - 1 mg tropicamide, 3 mg tropicamide, 0 mg tropicamide, 0.3 mg tropicamide
  Interventions: Drug: 0.3 mg tropicamide; Drug: 1 mg tropicamide; Drug: 3 mg tropicamide; Drug: 0 mg tropicamide
- Tropicamide 3 mg (Experimental): subject received (blinded) each of the 4 drug doses at different visits - 3 mg tropicamide, 0 mg tropicamide, 0.3 mg tropicamide, 1 mg tropicamide
  Interventions: Drug: 0.3 mg tropicamide; Drug: 1 mg tropicamide; Drug: 3 mg tropicamide; Drug: 0 mg tropicamide

INTERVENTIONS:
Drug: 0.3 mg tropicamide — 0.3 mg tropicamide in intra-oral thin film
  Other Names: NH004
Drug: 1 mg tropicamide — 1 mg tropicamide in intra-oral thin film
  Other Names: NH004
Drug: 3 mg tropicamide — 3 mg tropicamide in intra-oral thin film
  Other Names: NH004
Drug: 0 mg tropicamide — 0 mg tropicamide (placebo) in intra-oral thin film
  Other Names: NH004 (placebo)

SUMMARY:
The primary goal of the study is to evaluate the safety and potential efficacy of intra-oral dissolvable NH004 films to improve the short-term symptoms of sialorrhea (drooling) in Parkinson's disease (PD) patients.

DETAILED DESCRIPTION:
NH004 contains the anticholinergic agent tropicamide and is delivered in a convenient product form (intra-oral dissolvable thin films) designed for the management of sialorrhea. This study is a double blind, placebo-controlled, crossover study of the safety and potential efficacy of three doses of of NH004 films for the short-term relief of the symptoms of sialorrhea in Parkinson's disease patients.

A total of up to 36 Parkinson's disease patients will be enrolled in the study in two Phases. Phase A will include 12 patients and Phase B up to 24 patients. There will be an interim analysis after conclusion of Phase A. In both phases patients will be randomized into one of four groups. Each group will have a distinctive sequence for receiving intra-oral dissolvable films of 0.3 mg, 1 mg, 3 mg of NH004, or placebo during four visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with idiopathic Parkinson's disease, according to the United Kingdom Brain Bank criteria.
2. Patients complaining of drooling, with a score of at least 3 in the FLENI Sialorrhea scale.
3. Patient is between 50 and 80 years of age, inclusive.
4. Male or non-pregnant female. Females of child-bearing potential will be required to have undergone a pregnancy test with negative results prior to entry to the study and agree to use contraceptive measures for the duration of the study.
5. Patients must have used the same medication and dose for PD for the last month. No changes in the medication for PD are expected during the study.
6. Patients who can reasonable be expected to be on "on-state" for the duration of the testing procedures.
7. Patients who have a stable response to levodopa for PD.

Exclusion Criteria:

1. Pregnant women or women who may become pregnant.
2. Patients with a diagnosis of depression, schizophrenia or with obvious symptoms of these diseases.
3. Patients with Mini-Mental State Examination (MMSE) score equal to or lower than 26.
4. Patients who are receiving the following drugs: tricyclic antidepressants, Monoamine Oxidase Inhibitors (MAOI's), neuroleptics (antipsychotics), or anticholinergics.
5. Patients who have taken any of the drugs mentioned in exclusion criteria number 4 within the last week.
6. Patients with hypersensitivity to atropine or other anticholinergic drugs.
7. Patients who have experienced adverse effects as a result of taking anticholinergic drugs.
8. Patients taking hypnotic or other sleep inducing drugs.
9. Patients with severe urinary or gastrointestinal symptoms.
10. Patients with significant dental/oral pathology.
11. Patients with severe dysautonomia.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elkan R Gamzu, PhD, Principal Investigator — NeuroHealing Pharmaceuticals Inc.; Marcelo Merello, MD, PhD, Principal Investigator — FLENI Hospital, Argentina
Locations (1):
- FLENI Hospital, Buenos Aires, Argentina

REFERENCES:
- [Result] Lloret SP, Nano G, Carrosella A, Gamzu E, Merello M. A double-blind, placebo-controlled, randomized, crossover pilot study of the safety and efficacy of multiple doses of intra-oral tropicamide films for the short-term relief of sialorrhea symptoms in Parkinson's disease patients. J Neurol Sci. 2011 Nov 15;310(1-2):248-50. doi: 10.1016/j.jns.2011.05.021. Epub 2011 Jun 1. PMID 21636098

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four interventions, subjects were randomly assigned to one of 16 sequences.
Groups:
- All Participants: subjects randomly received (blinded) each of the 4 doses at different visits - 0 mg, 0.3 mg, 1mg, 3 mg Drug: Tropicamide
Period: Overall Study
Arm/Group | All Participants
Started | 19
Placebo | 19
0.3 mg Tropicamide | 19
1 mg Tropicamide | 19
3 mg Tropicamide | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This study was a double-blind, randomized, placebo controlled, two-phased, Latin-square crossover study. Subjects received three single-doses of tropicamide or placebo in random order, with a 7-day washout period.
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Region of Enrollment [Number; unit: participants]
  Argentina | 19

OUTCOME MEASURES:

1. Primary Outcome: Sialorrhea Visual Analogue Scale (VAS)
Description: Saliva buccal assessment was evaluated by an VAS scale before, and 15, 30, 45, 60, 90, and 120 min after treatment administration. Subjects were asked to rate how much saliva they perceived in their buccal cavity on an unmarked 0 to 10 cm line, higher scores meaning greater perceived buccal saliva levels.
Time Frame: Before and 120 min after treatment administration
Measure: Mean (Standard Deviation); unit: cm on VAS
Groups:
- Tropicamide - Placebo: Each subject randomly received blinded a placebo thin film containing no active drug ingredient
- Tropicamide - 0.3 mg: Each subject randomly received blinded a thin film containing 0.3 mg active drug ingredient
- Tropicamide - 1 mg: Each subject randomly received blinded a thin film containing 1 mg active drug ingredient
- Tropicamide 3 mg: Each subject randomly received blinded a thin film containing 3 mg active drug ingredient
Arm/Group | Tropicamide - Placebo | Tropicamide - 0.3 mg | Tropicamide - 1 mg | Tropicamide 3 mg
Number analyzed (Participants) | 19 | 19 | 19 | 19
cm on VAS | -0.55 (0.54) | -1.08 (0.54) | -1.53 (0.52) | -0.81 (0.51)
Statistical Analysis 1: Comparison: Tropicamide - Placebo vs Tropicamide - 0.3 mg vs Tropicamide - 1 mg vs Tropicamide 3 mg; Primary outcome was analyzed by a mixed-effects ANOVA model employing "subject" as a random factor as well as "visit" and "treatment" as fixed factors. Intention-to-treat (ITT) sample was analyzed. Unweighted means and their 95% Confidence Interval (CI) are reported, which represent treatment group means adjusted for the effect of visit and removing the intra-subject variability. For all analyses, significance level was set at 5%; Test type: Superiority or Other; p = 0.6, ANOVA

2. Secondary Outcome: Percentage Change in Saliva Volume
Description: Saliva volume was measured at baseline and 75 minutes after treatment administration. Volumes were measured by using cotton rolls placed near each Stenton duct and below the tongue for 5 minutes; cotton rolls were centrifuged and the volume of saliva determined.
Time Frame: Before and 75 minutes after treatment administration
Population: Percentage saliva volume change was determined in the last seven (7) patients enrolled.
Measure: Median (95% Confidence Interval); unit: percentage change of saliva volume
Arm/Group | Tropicamide - Placebo | Tropicamide - 0.3 mg | Tropicamide - 1 mg | Tropicamide 3 mg
Number analyzed (Participants) | 7 | 7 | 7 | 7
percentage change of saliva volume | -5 [-27 to 17] | -27 [-48 to -6] | -33 [-60 to -7] | -20 [-33 to -7]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- All Participants: subjects received (blinded) each of the 4 doses at different visits - 0 mg, 0.3 mg, 1mg, 3 mg Drug: Tropicamide
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less